CLINICAL TRIAL: NCT00375089
Title: Prader-Willi Syndrome and Early-onset Morbid Obesity Natural History Clinical Protocol
Brief Title: Characteristics of Prader-Willi Syndrome and Early-onset Morbid Obesity
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: RDCRN 5202; U54HD061222 (NIH); ARP 5202 (Other: RDCRN)
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Prader-Willi Syndrome; Obesity
Keywords: Early-onset Morbid Obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for both DNA and RNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Individuals with Prader-Willi syndrome.
  Interventions: Other: Group 1
- Group 2: Individuals with Early-onset Morbid Obesity
  Interventions: Other: Group 2

INTERVENTIONS:
Other: Group 1 — Individuals with Prader-Willi syndrome. Monitoring every 6 months.
  Other Names: Prader-Willi syndrome; PWS
  Groups: Group 1
Other: Group 2 — Individuals with Early-onset Morbid Obesity.
  Other Names: PWS
  Groups: Group 2

SUMMARY:
Prader-Willi syndrome (PWS) is a rare genetic disorder that affects about 1 in 14,000 people in the United States. As the most commonly identified genetic cause of obesity, PWS is often confused with Early-onset Morbid Obesity (EMO). Individuals with EMO show some signs of PWS, but clinically do not have PWS. The purpose of this study is to evaluate the clinical features and genetic basis of PWS and EMO, and to determine how these conditions affect a person throughout a lifetime.

DETAILED DESCRIPTION:
PWS is a complex neurobehavioral syndrome. Clinical features include obesity, increased appetite, low muscle tone, cognitive impairment, distinct behavioral features, hypogonadism, and neonatal failure-to-thrive. It is the most commonly recognized genetic cause of obesity; however, many obese children do not in fact have PWS. These individuals are therefore diagnosed with EMO, a condition that shares features with PWS. The development of new advances and strategies for treating PWS and EMO requires a thorough understanding of the conditions at both the clinical and molecular levels. One goal of this study is to collect long-term data on individuals with PWS and EMO in order to gain a better understanding of the natural progression of the conditions, from the neonatal period well into adulthood. Specific to PWS, this study will establish a genotype-phenotype correlation among the different sub-types and will evaluate the effects of growth hormone treatment on disease progression. Lastly, the study will compare PWS with EMO in terms of clinical features and genetic basis.

Participation in this natural history study will entail an initial evaluation, followed by yearly study visits until the age of 3 and then every 2 years thereafter. Each study visit will last between 3 and 4 hours, and will include a physical exam (including a DEXA scan to determine body composition), psychological testing, an interview with the study physician, and an evaluation of the participant's diet history. In addition, blood tests will be completed for genetic testing and photos will be taken to evaluate disease progression. Cognitive and behavioral assessments will also be conducted and will last between 10 and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolling in the Prader-Willi syndrome group will have a confirmed diagnosis of Prader-Willi syndrome, as confirmed by molecular and cytogenetic testing
* Individuals enrolling in the Early-onset Morbid Obesity group will have a documented medical history of their weight exceeding 150% of the ideal body weight or a body mass index greater than 97% before the age of 4 years; they will also be under the age of 30 years.

Exclusion Criteria:

* Known genetic, chromosomal, or hormonal cause of cognitive impairment other than Prader-Willi syndrome

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with Prader-Willi syndrome and Early-onset Morbid Obesity
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2006-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Phenotypic assessments of participants | until end of study
  phenotypic assessments will include cognitive level, behavioral analysis, physical features including body measurements and composition, co-morbidities (skin picking, psychiatric history, seizures, autistic behavior) medications required, and further comparison with the underlying molecular diagnosis.

SECONDARY OUTCOMES:
longitudinal pattern of progression | until end of study
  assessment of cognition, behavior and body composition. In addition the age that growth hormone treatment began in the PWS participants will be correlated with physical features, body composition, cognition, behavior, developmental milestones, pubertal issues, and the onset of nutritional phases.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Beaudet, MD, Study Chair — Baylor College of Medicine
Locations (4):
- United States (4):
  - University of California at Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Miller J, Kranzler J, Liu Y, Schmalfuss I, Theriaque DW, Shuster JJ, Hatfield A, Mueller OT, Goldstone AP, Sahoo T, Beaudet AL, Driscoll DJ. Neurocognitive findings in Prader-Willi syndrome and early-onset morbid obesity. J Pediatr. 2006 Aug;149(2):192-8. doi: 10.1016/j.jpeds.2006.04.013. PMID 16887432
- [Background] Miller JL, Couch JA, Schmalfuss I, He G, Liu Y, Driscoll DJ. Intracranial abnormalities detected by three-dimensional magnetic resonance imaging in Prader-Willi syndrome. Am J Med Genet A. 2007 Mar 1;143A(5):476-83. doi: 10.1002/ajmg.a.31508. PMID 17103438
- [Background] Butler MG. Management of obesity in Prader-Willi syndrome. Nat Clin Pract Endocrinol Metab. 2006 Nov;2(11):592-3. doi: 10.1038/ncpendmet0320. No abstract available. PMID 17082801
- [Background] Butler MG, Bittel DC, Kibiryeva N, Talebizadeh Z, Thompson T. Behavioral differences among subjects with Prader-Willi syndrome and type I or type II deletion and maternal disomy. Pediatrics. 2004 Mar;113(3 Pt 1):565-73. doi: 10.1542/peds.113.3.565. PMID 14993551
- [Background] Dykens E, Shah B. Psychiatric disorders in Prader-Willi syndrome: epidemiology and management. CNS Drugs. 2003;17(3):167-78. doi: 10.2165/00023210-200317030-00003. PMID 12617696
- [Background] Goldstone AP. Prader-Willi syndrome: advances in genetics, pathophysiology and treatment. Trends Endocrinol Metab. 2004 Jan-Feb;15(1):12-20. doi: 10.1016/j.tem.2003.11.003. PMID 14693421
- [Background] Miller J, Silverstein J, Shuster J, Driscoll DJ, Wagner M. Short-term effects of growth hormone on sleep abnormalities in Prader-Willi syndrome. J Clin Endocrinol Metab. 2006 Feb;91(2):413-7. doi: 10.1210/jc.2005-1279. Epub 2005 Nov 29. PMID 16317059
- [Background] Shapira NA, Lessig MC, He AG, James GA, Driscoll DJ, Liu Y. Satiety dysfunction in Prader-Willi syndrome demonstrated by fMRI. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):260-2. doi: 10.1136/jnnp.2004.039024. PMID 15654046
- [Background] Bittel DC, Butler MG. Prader-Willi syndrome: clinical genetics, cytogenetics and molecular biology. Expert Rev Mol Med. 2005 Jul 25;7(14):1-20. doi: 10.1017/S1462399405009531. PMID 16038620
- [Background] Holsen LM, Zarcone JR, Brooks WM, Butler MG, Thompson TI, Ahluwalia JS, Nollen NL, Savage CR. Neural mechanisms underlying hyperphagia in Prader-Willi syndrome. Obesity (Silver Spring). 2006 Jun;14(6):1028-37. doi: 10.1038/oby.2006.118. PMID 16861608
- [Background] Cassidy SB, Driscoll DJ. Prader-Willi syndrome. Eur J Hum Genet. 2009 Jan;17(1):3-13. doi: 10.1038/ejhg.2008.165. Epub 2008 Sep 10. PMID 18781185